CLINICAL TRIAL: NCT05565625
Title: A Single-Center, Clinical Study to Evaluate the Whitening Effect of Mineral Sunscreens in Multi-Cultural Skin Tones Thru Instrumentation Measurements, Imaging, and Self-Assessments
Brief Title: A Study to Evaluate the Whitening Effect of Mineral Sunscreens in Multi-Cultural Skin Tones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA004479; CCSSKA004479 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2022-09-15; First posted 2022-10-04 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sunscreen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunscreen (Experimental): Participants will receive two of six sunscreens (A, B, C, D, E, and F) at Visit 1 (Day 1) to apply to whole lower legs (1 sunscreen per lower leg), between the knee and ankle. Participant will then select one of the two sunscreens randomly assigned to lower legs and apply the selected sunscreen to full face. After lower legs and facial applications are completed, a trained designee will delineate six 4 centimeters (cm)*4 cm test sites on the participants' volar forearms (3 test sites per volar forearm). The six sunscreens will be randomly assigned to the six test sites at a dose of 2.00 +- 0.05 milligrams per centimeter square (mg/cm^2) using a 1cc tuberculin syringe (without a needle) and a clean finger cot for approximately 20 to 50 seconds and applied by a trained designee.
  Interventions: Other: Sunscreen A; Other: Sunscreen B; Other: Sunscreen C; Other: Sunscreen D; Other: Sunscreen E; Other: Sunscreen F

INTERVENTIONS:
Other: Sunscreen A — Participants will topically apply Sunscreen A at Visit 1.
Other: Sunscreen B — Participants will apply Sunscreen B at Visit 1.
Other: Sunscreen C — Participants will apply Sunscreen C at Visit 1.
Other: Sunscreen D — Participants will apply Sunscreen D at Visit 1.
Other: Sunscreen E — Participants will apply Sunscreen E at Visit 1.
Other: Sunscreen F — Participants will apply Sunscreen F at Visit 1.

SUMMARY:
The purpose of this study is to evaluate the whitening potential effect of different mineral sunscreens across multi-cultural skin tones through instrumentation, imaging, and self-assessment and also evaluate the relationship between self-perception and objective measurement of whitening.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported natural skin tone/skin color, targeting the following: skin tones "Pale/fair to light white" and "White to light beige" (n = 30 participants), skin tones "Beige to light tan/light olive" and "Medium tan/medium olive to light brown" (n = 30 participants), and Skin tones "Medium brown to dark brown" and "darkest brown to darkest black" (n = 30 participants)
* Has a history of using or is a current user of sunscreens
* Generally, in good health based on medical history reported by the participants
* Able to read, write, speak, and understand English
* Individual has signed the consent for photograph release and informed consent document (ICD) including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products or ingredients in the ISMs
* Presents with a skin condition on the face, volar forearms, or lower legs that may confound the study results (example, psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer) or interfere with evaluations (example, excessive hair, tattoos, scarring, very uneven skin tone, sunburn, scratches/broken/compromised skin)
* Has shaved or used any hair removal method on lower legs or volar forearms within 24 hours of Visit 1
* Has a history of a confirmed or suspected coronavirus disease 2019 (COVID-19) infection within 30 days prior to the study visit
* Within 14 days prior to Visit 1, has been in close contact (exposure within 6 feet for a cumulative time of 15 minutes or more over a 24-hour period) with anyone who has been infected with COVID-19
* Is under a COVID-19 isolation/quarantine order
* Has experienced any of the following self-reported symptoms of COVID-19 within 2 weeks prior to the study visit: unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, or chest pain/tightness; temperature greater than or equal to (>=) 37.5 degrees celsius (C)/99.5 degrees fahrenheit (F), measured; use of fever or pain reducers within 2 days prior to the study visit
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an adverse event (AE) or confound the study results, including: Immunosuppressive or steroidal drugs within 2 months before Visit 1; non-steroidal anti-inflammatory drugs within 5 days before Visit 1; antihistamines within 1 week before Visit 1
* Is self-reported to be pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other clinical study or has participated in any product-use study within 14 days prior to Visit 1
* Is an employee/contractor or immediate family member of the principle investigator (PI), study site, or sponsor

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Instrumentation | Visit 1 (Day 1)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through instrumentation (SkinSkan measurements) will be reported. SkinSkan is a non-invasive diagnostic tool that uses an optical fiber probe to collect the fluorescence signal from skin after excitation light is delivered through the same fiber probe.
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Imaging | Visit 1 (Day 1)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through imaging (facial and vocal forearms) will be reported. Image analysis will be done by using the Matlab software. A small region of interest (ROI) will be defined on the gray standard, and five regions on the face (forehead, nose, chin, left cheek, and right cheek) and the test regions on the volar forearms. The average RGB (red, green, and blue) values from these ROI will be extracted from the images. The RGB values from the gray standard will be used to calculate the correction factors per image based on the gray standard's target RGB values. Matlab will be used to convert the corrected RGB values to the LAB values. Skin whitening defined as the change in L* values pre and post product application. L* value is defined as lightness in LAB color space. High L* value corresponds to whiter color while low L* value corresponds to blacker color.
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Self-assessment | Visit 1 (Day 1)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through self-assessment will be reported via self-assessment questionnaire (Part B). This questionnaire rank whitening potential after application of the sunscreen product to the designated test areas on both inner forearms in order of least whitening (1) to most whitening (6).
Relationship Between Self-assessment and Instrumentation | Visit 1 (Day 1)
  Relationship between self-assessment and instrumentation (sunscreen product) will be reported via self-assessment questionnaire (Part A) which include the question about 'how much did you like or dislike the appearance of the sunscreen product on your skin' rated on a 5-point likert scale where 1 indicates "disliked it very much", 2 indicates "disliked it somewhat", 3 indicates "neither liked or disliked it", 4 indicates "liked it somewhat" and 5 indicates "liked it very much".

SECONDARY OUTCOMES:
Rate of Usage Versus Whitening Effect from a Sunscreen | Visit 1 (Day 1)
  Whitening effect from a sunscreen that impacts participant application behavior and ultimately their sun protection will be reported. This is being determined by correlation of the self-application dosage (milligrams per centimeter square [mg/cm^2]) per treatment area versus measured whitening effect (delta L*).
Skin Reflectance Before and After Sunscreen Applications as Assessed by SkinSkan Instrument | Visit 1 (Day 1)
  Skin reflectance will be assessed by SkinSkan instrument. SkinSkan instrument is a non-invasive diagnostic tool that uses an optical fiber probe to collect the signal from skin after excitation light is delivered through the same fiber probe. The spectra acquired at post sunscreen application and baseline for each site will be used to calculate Sun Protection Factor (SPF) following published Hybrid Diffuse Reflectance Spectroscopy (HDRS) method. Four replicates of spectra will be averaged to produce mean intensity of reflectance at baseline and sunscreen covered skin. Thus, each site measurement will produce one SPF level.

CONTACTS AND LOCATIONS:
Overall Officials: David Wrone, M.D., FAAD, Principal Investigator — Validated Claim Support (VCS)
Locations (1):
- Validated Claim Support (VCS), Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] U.S. Census Bureau. (n.d.). About race. Retrieved July 27, 2021, from https://www.census.gov/topics/population/race/about.html
- [Background] U.S. Census Bureau. (n.d.). About the Hispanic population and its origin. Retrieved July 27, 2021, from https://www.census.gov/topics/population/hispanic-origin/about.html
- [Background] Wan S, Anderson RR, Parrish JA. Analytical modeling for the optical properties of the skin with in vitro and in vivo applications. Photochem Photobiol. 1981 Oct;34(4):493-9. doi: 10.1111/j.1751-1097.1981.tb09391.x. PMID 7312955
- [Background] Mark Ruzon (2021). RGB2Lab (https://www.mathworks.com/matlabcentral/fileexchange/24009-rgb2lab), MATLAB Central File Exchange. Retrieved November 29, 2021.
- [Background] Mosteller RD. Simplified calculation of body-surface area. N Engl J Med. 1987 Oct 22;317(17):1098. doi: 10.1056/NEJM198710223171717. No abstract available. PMID 3657876
- [Background] Murari A, Singh KN. Lund and Browder chart-modified versus original: a comparative study. Acute Crit Care. 2019 Nov;34(4):276-281. doi: 10.4266/acc.2019.00647. Epub 2019 Nov 29. PMID 31795625
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKA004479&attachmentIdentifier=803ed870-6959-4ce4-b25a-a19cecb6dc20&fileName=CCSSKA004479_CSR_Synopsis_English.pdf&versionIdentifier=